CLINICAL TRIAL: NCT02762474
Title: A Phase I/II Trial of Weekly Regimens of Nab-paclitaxel Plus Cispaltin Combined With Concurrent IMRT for Inoperable,Locally Advanced Esophageal Carcinoma
Brief Title: Trial of Concurrent Chemoradiotherapy for Locally Advanced Esophageal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESO20140703
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Cancer
Keywords: nab-paclitaxel; IMRT; esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nab-paclitaxel group (Experimental): Weekly Regimens of paclitaxel Plus Cispaltin Combined With Concurrent IMRT
  Interventions: Drug: nab-paclitaxel group

INTERVENTIONS:
Drug: nab-paclitaxel group — Weekly Regimens of Nab-paclitaxel Plus Cispaltin Combined With Concurrent IMRT

SUMMARY:
This trial is going to evaluate the efficacy and safety of IMRT / nab-TP chemotherapy for unresectable esophageal cancer, and to investigate the optimal concurrent chemotherapy regimen for local advanced and unresectable esophageal cancer patients.

DETAILED DESCRIPTION:
Esophageal carcinoma is the sixth leading cause of cancer-related mortality from cancer with 407000 deaths and the eighth most common cancer worldwide. Concurrent chemoradiotherapy remains the mainstay of treatment for locally advanced esophageal cancer. Paclitaxel combined with radiotherapy was high efficiency and achieved encouraging results. Compared with paclitaxel, nab-paclitaxel has a low toxicity, low allergy and the tolerance is better than paclitaxel. According to the pre-clinical results, investigators designed a prospective study, which is combined nab-paclitaxel and cisplatin with concurrent chemoradiotherapy for the patients with locally advanced esophageal cancer, and evaluated the tolerability and efficacy. we design enrolled 30 patients, the end point included toxicity, progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. inoperable locally advanced histologically confirmed esophageal cancer (T3N0M0-TxNxM1a（AJCC 2002)
2. ECOG performance status scale 0-1
3. at least 1 measurable target lesions
4. white blood count ≥ 3,500/mm3, absolute neutrophil count ≥ 1,500/mm3, platelet count ≥ 100,000/mm3, hemoglobin count ≥ 90 g/dL, serum bilirubin level < 1.5 of the upper limit of normal (ULN) for the institution, aspartate aminotransferase, alanine aminotransferase and alkaline phosphatase ≤ 2.5 ULN, serum albumin ≥ 30g/L, serum creatinine ≤ 1.5 ULN; and
5. normal cardiac function with no severe heart disease.

Exclusion Criteria:

1. history of esophagectomy
2. pregnancy or breast feeding
3. past history of other cancers except for cured non-melanoma skin cancer or cervical cancer;
4. concomitant treatment with other anticancer drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years
CTCAE 4.0 toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ping Wang, M. D., Principal Investigator — Tianjin Medical University Cancer Hospital
Locations (1):
- Department of Radiation Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided